CLINICAL TRIAL: NCT03092518
Title: Phase II Trial of Heated Intraperitoneal Chemotherapy and Gastrectomy for Gastric Cancer With Positive Peritoneal Cytology
Brief Title: Heated Intraperitoneal Chemotherapy and Gastrectomy for Gastric Cancer With Positive Peritoneal Cytology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeremy Davis, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170070; 17-C-0070
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Gastric Adenocarcinoma; Esophagogastric Junction; Gastric Cancer
Keywords: Surgical Resection; Progression Free Survival; Gastroesophageal junction (Siewert III) adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Surgical Procedures, Operative; Cisplatin; Mitomycin; sodium thiosulfate; Positron Emission Tomography Computed Tomography; Magnetic Resonance Imaging; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer (Experimental): Heated Intraperitoneal Chemotherapy (HIPEC) with gastrectomy
  Interventions: Procedure: Surgery; Drug: Cisplatin; Drug: Mitomycin C; Drug: Sodium Thiosulfate; Procedure: Tumor Biopsy; Diagnostic Test: CT C/A/P; Diagnostic Test: PET-CT; Diagnostic Test: MRI; Diagnostic Test: EKG

INTERVENTIONS:
Procedure: Surgery — Heated Intraperitoneal Chemotherapy (HIPEC) with gastrectomy using cisplatin, mitomycin C and sodium thiosulfate
Drug: Cisplatin — Cisplatin (90 mg/m^2) will be administered via circuit to the peritoneal cavity
  Other Names: Platinol
Drug: Mitomycin C — Mitomycin C 10 mg/m^2 will be administered via circuit to the peritoneal cavity
  Other Names: Mitosol; Mutamycin; Jelmyto
Drug: Sodium Thiosulfate — Sodium thiosulfate will be administered by continuous intravenous infusion starting immediately prior to the chemotherapy perfusion and continuing for a total of 12 hours.
  Other Names: Sodium Thiosulfate Anhydrous; Sodium Hyposulfite; Sodium Thiosulfate Crystal; Prismatic Rice
Procedure: Tumor Biopsy — At screening, baseline (if not done at screening) and operation (as clinically indicated).
Diagnostic Test: CT C/A/P — At screening, baseline (if not done at screening), post op care, post-discharge visits/follow-up, semi-annual follow-up and annual follow-up.
  Other Names: Computed Tomography of the chest, abdomen and pelvis
Diagnostic Test: PET-CT — At screening, baseline (if not done at screening), post op care, post-discharge visits/follow-up, semi-annual follow-up and annual follow-up.
  Other Names: Positron emission tomography - computed tomography
Diagnostic Test: MRI — If computed tomography (CT) contraindicated.
  Other Names: Magnetic Resonance Imaging
Diagnostic Test: EKG — At screening and baseline (if not done at screening).
  Other Names: Electrocardiogram

SUMMARY:
Background:

- Gastric cancer is a common and serious cancer. Standard treatment is chemotherapy drugs. Researchers want to see if a new treatment helps. It is surgical removal of the cancer and heated chemotherapy delivered to the abdominal cavity called Hyperthermic intraperitoneal chemotherapy (HIPEC).

Objective:

- To test if surgical removal of tumors plus heated intraperitoneal chemotherapy can improve survival in people with gastric cancers.

Eligibility:

- People ages 18 and older with gastric cancer who can have most tumors surgically removed

Design:

* Participants will be screened with:
* Medical history
* Physical exam
* Blood, urine, and heart tests
* Scans
* Tissue sample from previous surgery
* Endoscopy with biopsy: A tube with a camera goes through the mouth and into the stomach. It and takes a sample of stomach tissue. Participants may get medicine to make them drowsy.
* Laparoscopy: Small cuts are made in the abdomen. A thin tube with a light and camera is inserted into the abdomen. Participants sleep through the procedure.

Participants will stay in the hospital. They will have:

* Surgery to remove as many tumors as possible.
* HIPEC for 60 minutes: Two thin tubes are put into the abdomen. Two chemotherapy drugs are given through one tube. They are drained out through another at a temperature a few degrees above normal body temperature. Another drug is given in a vein.
* Recovery for 7-21 days: Participants will have tubes in their stomach and bladder and intravenous (IVs) for a few days. They will get pain medicine, IV fluids, antibiotics, and blood transfusions as needed.
* Participants will have visits every few months for 3 years, then one a year. Visits include physical exam, blood tests, and scans. They also include dietary assessment and questions.

DETAILED DESCRIPTION:
Background:

* An estimated 24,590 cases of gastric adenocarcinoma are diagnosed annually in the United States (U.S.).
* The peritoneal surface is a site of metastasis found often at time of diagnosis and is a common (40%) site of recurrence.
* Laparoscopy with peritoneal lavage and cytopathologic analysis is a staging modality that can identify a subset of patients with microscopic peritoneal metastasis prior to consideration for definitive surgical therapy.
* Intraperitoneal chemotherapy has been employed in advanced gastric cancers and as an adjuvant with an associated improvement in survival in systematic reviews.

Objectives:

- Determine the overall survival in patients with cytology-positive gastric cancer treated with Hyperthermic intraperitoneal chemotherapy (HIPEC) and gastrectomy.

Eligibility:

* Histologically confirmed adenocarcinoma of the stomach.
* Cytopathologic evidence of peritoneal carcinomatosis.
* Medically fit for systemic chemotherapy, HIPEC and gastrectomy.

Design:

- Single arm, Phase II study of HIPEC and gastrectomy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed gastric adenocarcinoma or gastroesophageal junction (Siewert I-III) adenocarcinoma confirmed by the Laboratory of Pathology, national Cancer Institute (NCI).
* Must have received systemic chemotherapy, minimum 3 months or maximum 6 months, prior to enrollment
* Systemic therapy should consist of at least fluoropyrimidine-based and/or platinum-based chemotherapy
* Trastuzumab may be added for human epidermal growth factor receptor 2 (HER2)-neu over-expressing cancers as clinically indicated
* Last dose of chemotherapy within 8 weeks of enrollment with recovery to Grade 1 from chemotherapy-related toxicities
* Documentation of chemotherapy administration must be obtained
* Subradiographic and/or cytopathologic evidence of peritoneal carcinomatosis found at staging laparoscopy.
* Documentation of cytopathologic diagnosis of malignant peritoneal cytology in the absence of disseminated peritoneal disease must be obtained. If cytologic analysis reveals atypical cells of undetermined significance, a repeat lavage with cytopathologic analysis will be performed and must demonstrate evidence of malignancy.
* Limited peritoneal involvement found at staging laparoscopy or on final pathology that is deemed completely resectable is permitted
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* Patients must have normal organ and marrow function as defined below:
* hemoglobin > 8.0 g/dL
* absolute neutrophil count greater than or equal to 1,000/mcL
* platelets greater than or equal to100,000/mcL
* total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)Serum glutamic-oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT)Serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 X institutional upper limit of normal
* creatinine < 1.5 mg/dl
* estimated glomerular filtration rate (GFR) (creatinine clearance) greater than or equal to 60 mL/min/1.73 m^2.
* Physiologically able to undergo heated intraperitoneal chemotherapy (HIPEC) and gastrectomy
* No history of malignancy within 2 years of enrollment except for basal cell carcinoma of the skin, squamous cell skin cancer or carcinoma in situ of the cervix.
* Ability of subject to understand and the willingness to sign a written informed consent document
* Previous exploratory laparotomy or laparoscopy with tissue biopsy or peritoneal lavage is permitted.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Subjects must agree to co-enrollment on the tissue collection protocol 13C0176, Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors.

EXCLUSION CRITERIA:

* Patients who are receiving any investigational agents
* Disseminated extra-peritoneal or solid organ metastases
* Includes carcinomatosis associated with clinically or radiographically evident ascites (greater than 500cc)

  --Excludes greater omentum and ovarian metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because HIPEC and gastrectomy have not been studied in pregnant women and has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infant's secondary to treatment of the mother with HIPEC and gastrectomy, breastfeeding should be discontinued if the mother is treated on this study.
* Human immunodeficiency virus (HIV)-positive patients may be considered for this study only after consultation with a National Institute of Allergy and Infectious Diseases (NIAID) physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy L Davis, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Hartgrink HH, Putter H, Klein Kranenbarg E, Bonenkamp JJ, van de Velde CJ; Dutch Gastric Cancer Group. Value of palliative resection in gastric cancer. Br J Surg. 2002 Nov;89(11):1438-43. doi: 10.1046/j.1365-2168.2002.02220.x. PMID 12390389
- [Background] Mezhir JJ, Shah MA, Jacks LM, Brennan MF, Coit DG, Strong VE. Positive peritoneal cytology in patients with gastric cancer: natural history and outcome of 291 patients. Ann Surg Oncol. 2010 Dec;17(12):3173-80. doi: 10.1245/s10434-010-1183-0. Epub 2010 Jun 29. PMID 20585870
- [Background] Kang YK, Yook JH, Chang HM, Ryu MH, Yoo C, Zang DY, Lee JL, Kim TW, Yang DH, Jang SJ, Park YS, Lee YJ, Jung HY, Kim JH, Kim BS. Enhanced efficacy of postoperative adjuvant chemotherapy in advanced gastric cancer: results from a phase 3 randomized trial (AMC0101). Cancer Chemother Pharmacol. 2014 Jan;73(1):139-49. doi: 10.1007/s00280-013-2332-5. Epub 2013 Oct 27. PMID 24162381
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0070.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer: Heated Intraperitoneal Chemotherapy (HIPEC) with gastrectomy
  Surgery: Heated Intraperitoneal Chemotherapy (HIPEC) with gastrectomy using cisplatin, mitomycin C and sodium thiosulfate
  Cisplatin: Cisplatin (90 mg/m^2) will be administered via circuit to the peritoneal cavity
  Mitomycin C: Mitomycin C 10 mg/m^2 will be administered via circuit to the peritoneal cavity
  Sodium Thiosulfate: Sodium thiosulfate will be administered by continuous intravenous infusion starting immediately prior to the chemotherapy perfusion and continuing for a total of 12 hours.
  Tumor Biopsy: At screening, baseline (if not done at screening) and operation (as clinically indicated).
  Computed tomography chest/abdomen and pelvis (CT C/A/P): At screening, baseline (if not done at screening), post op care, post-discharge visits/follow-up, semi-annual follow-up and annual follow-up.
  Positron emission tomography-computed tomography (PET-CT): At screening, baseline (if not done at screening), post op care, post-discharge visits/follow-up, semi-annual follow-up and annual follow-up.
  Magnetic resonance imaging (MRI): If computed tomography (CT) contraindicated.
  Electrocardiogram (EKG): At screening and baseline (if not done at screening).
Period: Overall Study
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
Started | 27
Completed | 25
Not Completed | 2
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 22
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.81 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the median amount of time a participant survives after therapy.
Time Frame: 53.7 months
Population: 25/27 participants were analyzed because 2 were deemed ineligible.
Measure: Median (Full Range); unit: Months
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
Number analyzed (Participants) | 25
Months | 11.96 [5.42 to 19.71]

2. Secondary Outcome: Intraperitoneal Progression Free Survival (IPFS) at 6 Months, 12 Months and 18 Months
Description: Intraperitoneal progression free survival is defined as the median amount of time a participant survives from date of operation (hyperthermic intraperitoneal chemotherapy (HIPEC) and gastrectomy) without intraperitoneal disease progression after treatment. Intraperitoneal progression is defined as new, large volume ascites with or without associated peritoneal nodularity or thickening determined by radiographic imaging, cytopathology or histopathology.
Time Frame: 6 months, 12 months and 18 months
Population: 25/27 participants were analyzed because 2 were deemed ineligible.
Measure: Median (Full Range); unit: Months
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
Number analyzed (Participants) | 25
Months
  6 months | 0.9 [0.65 to 0.97]
  12 months | 0.83 [0.54 to 0.94]
  18 months | 0.83 [0.54 to 0.94]

3. Secondary Outcome: Extra-peritoneal Disease-free Survival
Description: Extra-peritoneal disease-free survival is defined as the median amount of time a participant survives from date of surgery to the date of first observation of progressive disease at sites other than the peritoneal surface (e.g., liver, intra-abdominal lymph nodes, abdominal wall soft tissues, and any other solid organs) determined by radiographic imaging (i.e., computed tomography, magnetic resonance imaging, and/or positron emission tomography).
Time Frame: 48.9 months
Population: 25/27 participants were analyzed because 2 were deemed ineligible.
Measure: Median (Full Range); unit: Months
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
Number analyzed (Participants) | 25
Months | 48.9 [0 to 48.9]

4. Secondary Outcome: Number of Treatment Related Serious and/or Non-serious Adverse Events by Type
Description: The number of treatment related serious and/or non-serious adverse events by type related to research treatments was assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Up to 1646 days
Population: 2/27 participants were deemed ineligible prior to treatment.
Measure: Number; unit: adverse events
Groups:
- Serious: All treatment related serious adverse events.
- Non-Serious: All treatment related non-serious adverse events.
Arm/Group | Serious | Non-Serious
Number analyzed (Participants) | 25 | 25
adverse events
  abdominal distension | 0 | 3
  Abdominal infection | 2 | 4
  Abdominal pain | 1 | 18
  Acidosis | 0 | 1
  Activated partial thromboplastin time prolonged | 0 | 2
  Acute kidney injury | 1 | 1
  Alanine aminotransferase increased | 0 | 15
  Alkaline phosphatase increased | 0 | 1
  Anemia | 12 | 69
  Anorexia | 0 | 2
  Anxiety | 0 | 2
  Ascites | 1 | 0
  Aspartate aminotransferase | 0 | 21
  Aspiration | 1 | 0
  Atelectasis | 0 | 2
  Atrial fibrillation | 4 | 0
  Atrial flutter | 1 | 0
  Back pain | 0 | 2
  Bladder perforation | 0 | 1
  Bloating | 0 | 3
  Blood bilirubin increased | 0 | 8
  CPK increased | 0 | 3
  Chest wall pain | 0 | 1
  Colitis | 0 | 1
  Confusion | 0 | 1
  Cough | 0 | 1
  Creatinine increased | 1 | 1
  Cystitis noninfective | 0 | 1
  Dehydration | 0 | 1
  Depressed level of consciousness | 1 | 0
  Depression | 0 | 2
  Diarrhea | 0 | 5
  Disseminated intravascular coagulation | 1 | 0
  Dizziness | 0 | 1
  Duodenal fistula | 1 | 0
  Dyspnea | 5 | 4
  Edema limbs | 0 | 6
  Esophageal anastomotic leak | 2 | 4
  Esophagitis | 1 | 0
  Fatigue | 0 | 3
  Fever | 1 | 12
  Gastrointestinal anastomotic leak | 1 | 0
  Headache | 0 | 1
  Hematuria | 0 | 1
  Hiccups | 0 | 5
  Hyperglycemia | 0 | 3
  Hyperkalemia | 1 | 1
  Hypernatremia | 0 | 2
  Hypertension | 2 | 8
  Hypoalbuminemia | 1 | 30
  Hypocalcemia | 0 | 7
  Hypokalemia | 1 | 4
  Hyponatremia | 2 | 3
  Hypophosphatemia | 0 | 48
  Hypotension | 4 | 15
  Hypothermia | 1 | 0
  Hypoxia | 1 | 1
  Infections and infestations-other | 1 | 0
  Insomnia | 0 | 2
  Intraoperative urinary injury | 0 | 1
  Lung infection | 3 | 1
  Lymphocyte count decreased | 0 | 44
  Malaise | 1 | 0
  Mediastinal infection | 1 | 0
  Metabolism and nutrition disorders other | 1 | 0
  Nausea | 0 | 11
  Neutrophil count decreased | 0 | 2
  Oral pain | 0 | 1
  Pain | 0 | 10
  Pain in extremity | 0 | 1
  Pericardial effusion | 0 | 1
  Platelet count decreased | 0 | 1
  Pleural effusion | 9 | 4
  Pleural infection | 2 | 0
  Pneumothorax | 0 | 1
  Productive cough | 0 | 1
  Renal and urinary disorders-other | 0 | 1
  Respiratory failure | 5 | 0
  Respiratory, thoracic and mediastinal disorders-other | 4 | 0
  Sepsis | 5 | 1
  Serum amylase increased | 0 | 1
  Sinus bradycardia | 1 | 0
  Sinus tachycardia | 3 | 11
  Small intestinal obstruction | 3 | 0
  Sore throat | 0 | 1
  Upper gastrointestinal hemorrhage | 2 | 1
  Urinary tract infection | 0 | 2
  Vaginal anastomotic leak | 0 | 1
  Vomiting | 0 | 8
  Weight loss | 2 | 6
  White blood cell decreased | 1 | 5

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Document adverse events from the first study intervention (pre-operation visit) through 30 days after removal from study treatment or until off-study, whichever comes first, approximately 365 days
Population: 25/27 participants were analyzed because 2 were deemed ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
Number analyzed (Participants) | 25
Participants | 23

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 53.7 months. Adverse Events monitored/assessed from the first study intervention (pre-operation visit) through 30 days after removal from study treatment or until off-study, whichever comes first, approximately 365 days.
Arm/Group | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer
All-Cause Mortality (participants affected / at risk) | 23/27
Serious Adverse Events (participants affected / at risk) | 10/27
Other Adverse Events (participants affected / at risk) | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer (N=27)
Abdominal infection (Infections and infestations) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (12)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (4)
Atrial flutter (Cardiac disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Duodenal fistula (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 2 (4)
Hypothermia (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, Bacteremia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (3)
Malaise (General disorders) | 1 (1)
Mediastinal infection (Infections and infestations) | 1 (1)
Metabolism and nutrition disorders - Other, Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Pleural infection (Infections and infestations) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Sepsis (Infections and infestations) | 4 (5)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heated Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer (N=27)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal infection (Infections and infestations) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 10 (19)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (15)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 22 (71)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 13 (21)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder perforation (Hepatobiliary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (8)
CPK increased (Investigations) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema limbs (General disorders) | 4 (6)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 4 (4)
Fatigue (General disorders) | 4 (4)
Fever (General disorders) | 8 (14)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (30)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (7)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 16 (48)
Hypotension (Vascular disorders) | 11 (16)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Intraoperative urinary injury (Injury, poisoning and procedural complications) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 14 (44)
Nausea (Gastrointestinal disorders) | 7 (12)
Neutrophil count decreased (Investigations) | 3 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal and urinary disorders - Other, Urinary Leak (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Serum amylase increased (Investigations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 8 (11)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vaginal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8)
Weight loss (Investigations) | 4 (6)
White blood cell decreased (Investigations) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03092518/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03092518/ICF_001.pdf